CLINICAL TRIAL: NCT03248154
Title: Burn Biofilm Infection in Adults and Children
Brief Title: Biofilm Infection in Adults and Children Burn Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: did not receive funding
Sponsor: Gayle Gordillo (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Gayle Gordillo, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00244
Record Dates: First submitted 2017-02-08; First posted 2017-08-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Thermal Burn; Wound
Keywords: Biofilm; Procellera
MeSH Terms: conditions — Wounds and Injuries

ARMS (3):
- Immunocompetent with 2-14% TBSA (No Intervention): Immunocompetent with 2-14% TBSA thermal burn subjects. Does biofilm infection result in conversion of partial-thickness burn wounds to full-thickness?
- Immunocompromised with >=20% TBSA (Experimental): Immunocompromised patients with large thermal burn >=20% TBSA. Higher bacterial burden with biofilm infection will result in higher rates of graft loss. Does application of a wireless electroceutical dressing (Procellera) lower biofilm burden compared to burn subjects receiving standard of care therapy?
  Interventions: Device: Procellera
- Peripheral blood - all subjects (No Intervention): All subjects enrolled in arms 1 and 2. Do children have a more robust innate immune response to prevent biofilm infection?

INTERVENTIONS:
Device: Procellera — burn dressing
  Arms: Immunocompromised with >=20% TBSA

SUMMARY:
The objective of the study is to analyze the different implications (such as graft loss and conversion of indeterminate depth burns) of biofilm infections in burn patients. Additionally, it also aims at comparing children's resistance to biofilm infection at wound site than adults'. 300 subjects from 3 different age groups will be enrolled in 3 arms.

DETAILED DESCRIPTION:
Subjects will be recruited from three different age groups: 2-18 years old, 18-49 years old, and ≥ 50 years old. 150 patients will be enrolled in each age group for arms 1 and 2. Arm 3 consists of all patients enrolled in the study and involves drawing whole blood for analyzing cytokine response. Subjects will have at day 0, 3, 7, 14, 21, 28 +/- 2 days (as applicable until graft surgery occurs).At each study visit the following will be collected: burn wound data [Lund-Brower Chart, TBSA burn size, date of onset, length, width, area, depth of burn injury (as applicable), Standard of Care (SoC) treatment for burn] will be recorded, SoC labs since the onset of the burn wounds will be recorded (CBC w/ diff and glucose as applicable), digital imaging of the burn injury(s), Laser Doppler Imaging (LDI) will also be perfomed. Biopsies will be collected depending on the size of injury (4 from 2cm² burn size, to 10 from >8cm² burn size). Blister fluid will be collected by draining the fluid with a needle and syringe.Subjects in arm 2 will receive their Standard of Care (SoC) dressing prescribed by their provider or will receive the study dressing, 4x4 Procellera that will be applied to a specific area of the burn injury.

2 weeks after the grafting surgery, subjects will return for study visits at day 14, 21, 28 post-grafting where the following activities will be completed - burn wound data and medication review, digital image of the burn injury(s), LDI imaging, HUSD imaging, trans-epidermal water loss (TEWL) measurement. Whole blood will be collected.

Each subjects' medical chart will be followed for 3 months post completion of the study to identify patient outcomes (i.e. wound closure data, infection status/type, treatment status, surgical outcomes/complications - graft loss, patient death as applicable).

ELIGIBILITY:
Inclusion Criteria (Aim 3 is included in all criteria):

Aim 1 and 2:

* Ages 2 yrs. and older

Aim 1:

* Thermal burns with 2-14% total body surface area (TBSA) injury
* Patients present within 3 days from the time of thermal burn injury
* Diagnosed by burn surgeon as having deep partial thickness or indeterminate depth burn (defined as uncertainty between deep second degree or third degree burns)

Aim 2:

* Thermal burns with ≥20% TBSA

Exclusion Criteria (Aim 3 is included in all criteria):

Aim 1 and 2:

* Patients with chemical or electrical burns
* Pregnant women
* Patient/legal guardian/or next of kin unable to consent

Aim 1:

* Immunosuppressed
* Taking immune modifying medications
* Patients requiring >72 hrs. hospital stay
* Harmonic Ultrasound & Doppler Imaging (HUSD) will be used to exclude burn wounds with thrombosed vessels at initial presentation

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Detection of biofilm infection in burns | 4 weeks
  Tissue biopsies will be tested for presence of bacteria using SEM and culture.

SECONDARY OUTCOMES:
Assessing graft loss as a result of biofilm infection | 4 weeks post grafting surgery
  TEWL measurement (g/square meter/h) as an indicator of lost barrier function
Burn depth measurement | 4 weeks
  Harmonic Ultrasound & Doppler (HUSD) imaging will provide tissue depth expressed in relevant unit

OTHER OUTCOMES:
Examining children vs adults for biofilm resistance | 2 weeks post grafting surgery
  TNF-a measurement through cytokine assay (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle M Gordillo, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - University Hospital East, Columbus, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - The Ohio State University/Ohio State University Wexner Medical Center, Columbus, Ohio
  - Martha Morehouse Medical Plaza 2050 Kenny Road, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No